CLINICAL TRIAL: NCT06632860
Title: a Novel Dual-Targeting Molecular Probe TATE-RGD for the Diagnostic Integration of SSTR2 and αvβ3 Positive Tumors
Brief Title: A Dual-targeting Tracer TATE-RGD for the Diagnosis of SSTR- and RGD- Positive Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhaohui Zhu, prof., Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-TR-DTC
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2024-10

CONDITIONS: Iodine-resistant Thyroid Cancer; Meningioma; NETs
MeSH Terms: conditions — Meningioma | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: 68Ga-TATE-RGD PET/ CT scan (Experimental): About 30 patients with positive expression of somatostatin receptor SSTR2 and integrin receptor αvβ3 were included for PET imaging.
  Interventions: Drug: 68Ga-TATE-RGD; Drug: 18-FDG

INTERVENTIONS:
Drug: 68Ga-TATE-RGD — Intravenous injection of 68Ga-TATE-RGD with the dosage of 1.8-2.2 MBq (0.05-0.06 mCi)/kg. Tracer doses will be used to image lesions of by dual-targeted postive cancers PET/CT.
Drug: 18-FDG — Intravenous injection of 18F-FDG with the dosage of 1.8-2.2 MBq(0.12-0.15mCi/kg). Tracer doses will be used to lesions therapy of dual-targeted postive cancers by SPECT/CT.

SUMMARY:
The US FDA approved a targeted somatostatin receptor 2 imaging agent, 68Ga-DOTATATE, in 2016. It has higher uptake in small cell lung cancer, pulmonary carcinoid, and medullary thyroid cancer. Integrin αvβ3 is highly expressed in some tumor cells and new blood vessels, making it an ideal target for targeted diagnosis and treatment of tumors and tumor vessels.68Ga-labeled DOTA-TATE-RGD is a new type of tumor-specific imaging agent developed by researchers based on the above foundation, which is used for targeted diagnosis and internal radiation therapy for patients with SSTR2 and αvβ3 positive tumors.

DETAILED DESCRIPTION:
This research has conducted extensive studies on the treatment of neuroendocrine tumors with 177Lu-EB-TATE and the treatment of FAP-expressing tumors with 177Lu-EB-FAPI. The same protocol had demonstrated 68Ga-TATE-RGD showed an increasing TBR, suggesting the tracer kinetic advantage of TATE-RGD. Compared to the single-target tracer DOTATATE, the dual-target TATE-RGD probe has a clear advantage in detecting NETs liver metastases, and it can be explored for potential therapeutic uses in future studies and used for related companion diagnostics in targeted radiolabeling therapy (RLT), which has been published in the 1st-impact factor journal European Journal of Nuclear Medicine and Medical Imaging (IF: 9.6), performing a small-dose diagnostic PET imaging with the same tracer.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed various cancer patients;
* 68Ga-TATE-RGD and 18F-FDG PET/CT within a week;
* signed written consent.

Exclusion Criteria:

* known allergy against TATE-RGD;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Tumor detection rate | through study completion, an average of half-year
  comparing the number of tumor detected by 68Ga-TATE-RGD and18F-FDG PET/CT

SECONDARY OUTCOMES:
standardized uptake value (SUV) of tumor | through study completion, an average of half-year
  comparing the SUVmax of tumor derived from 68Ga-TATE-RGD and 18F-FDG PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China